CLINICAL TRIAL: NCT00793611
Title: Hypnotherapy for Treatment of Overactive Bladder: A Feasibility Study
Brief Title: Hypnotherapy for Treatment of Overactive Bladder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Principal Investigator, Yuko Komesu, Assistant Professor Ob-Gyn University of new Mexico, University of New Mexico
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 08-102
Record Dates: First submitted 2008-10-06; First posted 2008-11-19 (Estimated); Results first posted 2011-10-28 (Estimated); Last update posted 2017-10-09 (Actual); Status verified 2017-09

CONDITIONS: Overactive Bladder
Keywords: Overactive Bladder; Hypnotherapy
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Behavior Therapy; Hypnosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Behavioral therapy (Active Comparator): "Behavioral Therapy standard of care (which consists of bladder drills, voiding diaries, timed voiding and pelvic floor exercises)"
  Interventions: Behavioral: Behavioral therapy standard of care
- hypnotherapy (Experimental): patients will receive 3 hypnotherapy sessions in addition to usual behavioral treatments for overactive bladder
  Interventions: Behavioral: Behavioral therapy standard of care; Other: hypnotherapy

INTERVENTIONS:
Behavioral: Behavioral therapy standard of care — controls will receive usual interventions for overactive bladder: voiding diary, bladder drills, pelvic floor exercises
  Other Names: behavioral treatment; pelvic floor exercise; bladder drills
Other: hypnotherapy — Patients will receive 3 hypnotherapy sessions in addition to usual behavioral treatment of overactive bladder
  Other Names: hypnosis
  Arms: hypnotherapy

SUMMARY:
The investigators purpose is to perform a pilot study evaluating the efficacy in hypnotherapy in treating women with Overactive Bladder Symptoms (urinary urgency symptoms and urinary frequency). Approximately half the women in the study will receive "standard care" (performing a voiding diary, Pelvic Floor exercises, and timed voiding) and the other half will receive "standard care" and 3 hypnotherapy sessions. The investigators will compare the groups using a validated overactive bladder questionnaire and compare voiding diaries to evaluate urinary frequency at the end of the sessions/study completion.

DETAILED DESCRIPTION:
Experimental Design and Methods:

i) This is a feasibility study (prior to performing a larger randomized controlled trial at a later date) evaluating whether hypnotherapy effectively treats Overactive Bladder (OAB). Ultimately, for the larger study, in order to find a 20% difference between the hypnotherapy group and controls, we will need to evaluate a total of approximately 66-70 women to find a 20% difference between groups, assuming 80% power and P=0.05. However, the purpose of this pilot study is to evaluate the feasibility of the larger study and determine the appropriate control intervention and outcomes. We plan to evaluate approximately ten subjects (approximately twenty overall) in both the control and hypnotherapy groups.

ii) Patients OAB will be offered entry into the study. a) Inclusion criteria: women experiencing 8 voids/day and an OAB Awareness tool score greater than 8. b) Exclusion criteria: males (since we do not care for males in the gynecology clinic), non-English speakers, pregnant women, women younger than 18 years old, incarcerated women, women with a history of bipolar disorder or schizophrenia, women unwilling to undergo hypnotherapy iii) Informed consent will be obtained. iv) Prior to receiving interventions, patients will be administered the OAB-q & instructed to keep a 3 day voiding diary. If the patient has not had a pelvic exam in the urogynecology clinic within the last year, a pelvic exam will be performed.

v) The usual standard treatments for OAB include pelvic floor exercise, voiding diaries, bladder drills (increasing time between voids), and anti-cholinergic medications. The control group will be offered any or all of our standard treatments, including Behavioral treatment (review of voiding diaries and instruction regarding behavioral changes). Both groups will be allowed to continue current OAB medications but asked not to start new medications. The hypnotherapy group will also be offered any or all of our standard treatments, but they will be given the option of receiving hypnotherapy in addition to the usual treatments.

vi) Hypnotherapy sessions: Dr. Sapien will conduct 3 hypnotherapy session to women randomized to the hypnotherapy group. These sessions will occur approximately every1-2 weeks over approximately a time span of 6-8 weeks. The sessions will last 60-90 minutes. Session #1) Explain hypnotherapy and practice suggestion therapy; Session #2) address emotions around OAB and life impact, visualization of pelvic floor exercise mechanics, teach self hypnosis; Session #3) address emotions, further practice on exercises and self-hypnosis vii) Blinding of Investigators and Allocation Concealment: Randomization will be performed by the CTSC using computer generated allocation. Only the CTSC personnel will know the assignment schema. Researchers will not know the group assignments. A research nurse otherwise uninvolved in the study will place the group assignments in serially numbered, opaque envelopes. Once subjects sign consents they will receive an opaque envelop assigning them to the Behavioral Therapy or Hypnotherapy group. The individual responsible for data collection and data entry will not know the group assignment until the end of the study when the assignment code is broken.

VI. Human Subjects:

i) See inclusion & exclusion criteria described previously. Children, prisoners and mentally ill or disabled subjects will be excluded from our study. Women who are pre-menopausal and who are not using contraception and have missed a menstrual period will be offered a pregnancy test in the clinic, as is the standard of care in the gynecology clinic. Pregnancy is an exclusion criteria for study participation.Women evaluated in the Gynecology Clinic at the University of New Mexico will be offered participation in the study.

ii) Women will be offered study participation in a private setting at their gynecology visit if have the symptoms of OAB noted previously (V.ii).The study will be described verbally and they will receive a copy of the consent form to read. They will be given the option of taking the consent home to have time to consider whether they would like to participate. If the patient wishes more time to consider whether she would like to participate, she will be asked whether she would agree to phone follow-up by a study investigator. If she agrees, she will have phone follow-up at least 24 hours after her clinic visit. If the patient expresses interest in participating in the study, she will then return to sign her consent with a study investigator. All patients will be reassured that declining study participation will have no effect on the care that they receive iii) Potential Risks of Hypnotherapy: Potential Risks of Hypnotherapy: Risks of hypnotherapy are minimal. Hypnosis is a natural state of mind in which the subconscious is accessed and utilized to make a positive impact. Although, in the 1980 false memory syndrome was described with the use of hypnotherapy in child abuse survivors, the current practice of hypnotherapy uses a much different approach to this therapeutic application. Current practice includes open-ended lines of questioning as opposed to suggestive or leading lines of questioning utilized with these victims.

Risks will be minimized by using open-ended lines of questioning for all hypnotherapy sessions (see above). For this study the hypnotherapist is also a physician, therefore physician-patient confidentiality guidelines are in place. Subjects will be asked to contact the PI if they believe that they are suffering from a psychological burden which has occurred from their involvement in the study.

It is highly unlikely that this study would be terminated, as the risks to participants are minimal. However, in the unlikely circumstance that a large number of hypnotherapy subjects complain of severe psychologic or physical discomfort with their hypnotherapy sessions (despite incorporation of relaxation techniques in the sessions), the study would be terminated. Subject case discussion will be conducted by the research team in a private setting

Potential Risks to Control Group: The control group will be offered standard care for treatment of OAB and will not be exposed to any greater risk than usual for OAB treatments iv) Potential Benefits of Hypnotherapy: Alleviating or diminishing symptoms of frequent urinary, urinary urgency and urine leakage.

v)Safety Oversite: The investigators will meet approximately monthly to review study progress and subject issues/complaints. The subjects will have follow-up with either phone or in-person contact with the hypnotherapist or CTSC personnel. If major events, though unlikely, occur, they will be reviewed with appropriate CTSC and HRRC personnel.

vi) After the study is finished, the patients in the control group have the option of undergoing an approx. 20 minute relaxation hypnotherapy session with Dr. Sapien.

ELIGIBILITY:
Inclusion Criteria:

* More than 8 voids/day
* Score > 8 on OABq questionnaire
* English speaking

Exclusion Criteria:

* Pregnancy
* Less than 18 years old
* History of Schizophrenia or Bipolar Disorder

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-11; Primary Completion 2010-01 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yuko M Komesu, MD, Principal Investigator — University of New Mexico Health Sciences Center

REFERENCES:
- [Result] Freeman RM, Baxby K. Hypnotherapy for incontinence caused by the unstable detrusor. Br Med J (Clin Res Ed). 1982 Jun 19;284(6332):1831-4. doi: 10.1136/bmj.284.6332.1831. PMID 6805716

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients recruited from the Clinic. Study received IRB approval winter 2008 and recruitment occurred 2008-10.
Groups:
- Behavioral Therapy Standard Care: received 3 behavioral therapy session
- Hypnotherapy: received 3 sessions of behavioral therapy combined with hypnotherapy
Period: Overall Study
Arm/Group | Behavioral Therapy Standard Care | Hypnotherapy
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Behavioral Therapy Standard Care | Hypnotherapy | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.4 (7.4) | 51.1 (14) | 54 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Change in Overactive Bladder Symptoms (Based on OABqSF)
Description: Scale information; Score ranges for oab-qsf quality of life scores range from 13-78; 13=poor quality of life 78=good quality of life. We reported change scores, with larger negative numbers indicating greater improvement in quality of life scores.
Time Frame: baseline and approximately 6-12 weeks after study initiation
Population: ITT
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Behavioral Therapy Standard Care | Hypnotherapy
Number analyzed (Participants) | 10 | 10
units on a scale | -19 (24.9) | -33.4 (15.2)
Statistical Analysis 1: Comparison: Behavioral Therapy Standard Care vs Hypnotherapy; ITT between group differences in change scores compared for behavioral therapy and hypnotherapy groups. Power analysis: This is a pilot study underpowered find between group differences based on our power analysis(a 20% difference between groups would require 88 women, assuming 80% power and α=0.05 based on Freeman's study cited later). The purpose of this pilot study is to evaluate the feasibility of the larger study and determine the appropriate control intervention and outcomes; Test type: Superiority or Other; p = .07, t-test, 2 sided; 19 degrees of freedom; Mean Difference (Net) = .20

2. Secondary Outcome: Change in Voiding Frequency Based on Voiding Diary
Description: change in mean number of voids per 24 hours. Each participant recorded voiding frequency every 24 hours for 3 days at baseline and follow-up. A mean number of voids for every patient over 24 hours was calculated at baseline and follow-up.
Time Frame: baseline and 6-12 weeks after study initiation
Population: ITT change in mean number of voids/24 hours
Measure: Mean (Standard Deviation); unit: number of voids per 24 hours
Arm/Group | Behavioral Therapy Standard Care | Hypnotherapy
Number analyzed (Participants) | 10 | 10
number of voids per 24 hours | 1.4 (1.4) | 2.6 (2.0)
Statistical Analysis 1: Comparison: Behavioral Therapy Standard Care vs Hypnotherapy; intent to treat; Test type: Superiority or Other; p = .17, t-test, 2 sided

3. Secondary Outcome: Patient Global Impression of Improvement
Description: Outcome measure is only administered at follow-up and used following treatment in patients with urinary incontinence. Measure varies from 1 to 7 on a Likert scale. 1=very much better and 7=very much worse and 4=no change. Thus, lower numbers represent greater improvement.
Time Frame: 6-12 weeks after study initiation (@ completion of intervention)
Population: ITT
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Behavioral Therapy Standard Care | Hypnotherapy
Number analyzed (Participants) | 10 | 10
units on a scale | 3.4 (.97) | 2.15 (.3)
Statistical Analysis 1: Comparison: Behavioral Therapy Standard Care vs Hypnotherapy; intent to treat; Test type: Superiority or Other; p = .009, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Behavioral Therapy Standard Care | Hypnotherapy
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes